CLINICAL TRIAL: NCT05878067
Title: A Patient Experience Study With ABBV-444 for Symptom Relief and Tolerability
Brief Title: A Study to Assess Symptom Relief and Product Tolerability of ABBV-444 Drops in Adult Participants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P24-203
Record Dates: First submitted 2023-05-24; First posted 2023-05-26 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Dry Eye Syndrome
Keywords: Dry Eye Syndrome; ABBV-444
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ABBV-444 (Experimental): Participants will administer 1-2 drops of ABBV-444 in each eye as needed but minimally twice a day for 30 days.
  Interventions: Drug: ABBV-444

INTERVENTIONS:
Drug: ABBV-444 — Lubricant Eye drops

SUMMARY:
Dry Eye Disease (DED) is a condition where the tear film of the eye becomes unstable and along with ocular surface inflammation and damage leads to inadequate tear production and eye lubrication. This study will evaluate symptom relief and tolerability of ABBV-444 eye drops in adult participants.

ABBV-444 is being developed for the treatment of Dry Eye Disease (DED). This is a 30-day, open-label study to evaluate adult participant symptoms and tolerability of ABBV-444. Around 40 participants will be enrolled in 1 site in the United States.

Participants will receive 1-2 drops of ABBV-444 in each eye as needed but minimally twice a day for 30 days.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Had used artificial tears for dry eyes within the past year
* OSDI score of ≥ 18 and ≤ 65 (based upon a 0 to 100 scale) at Screening and Baseline Visits Three consecutive tear breakup time (TBUT) tests ≤ 10 seconds in at least 1 eye at Day -7 (screening)
* Grade 1 to 4 (modified National Eye Institute [NEI] Grid, score range = 0 to 5) staining in at least 1 area of the cornea (5 areas examined) or conjunctiva (6 areas examined) that was related to dry eye in at least 1 eye at both at Screening and Baseline Visits

Exclusion Criteria:

* Have uncontrolled severe systemic disease that, in the assessment of the investigator, would put safety of the participant at risk through participation, or which would prevent or confound protocol-specified assessments (e.g., hypertension and diabetes, Sjögren's syndrome, rheumatoid arthritis, systemic lupus erythematosus, immunodeficiency disease, etc.)
* Known allergy or sensitivity to the study products or their components
* Schirmer Test (with anesthesia) ≤ 2 mm in either eye at Screening Visit
* Participant anticipated contact lens wear during the study, or the participant had worn contact lenses in the last 3 months prior to Screening Visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-06-27 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Canyon City Eyecare /ID# 253652, Azusa, California, United States

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=P24-203

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 40 participants were enrolled and included in the intent-to-treat (ITT) population. The per-protocol (PP) population included 34 participants after excluding 4 participants who were deemed protocol deviations and 2 participants who discontinued the study. The per-protocol population was used for all efficacy measures.
Pre-assignment Details: Four participants were deemed protocol deviations following data entry and analysis because their baseline OSDI scores were outside the 18 to 65 inclusion range. The 4 participants were not included in the per protocol population.
Groups:
- ABBV-444: Participants administered 1-2 drops of ABBV-444 in each eye as needed but minimally twice a day for 30 days.
  ABBV-444: Lubricant Eye drops
Period: Overall Study
Arm/Group | ABBV-444
Started | 40
Completed | 38
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: ITT population: Includes all enrolled participants who received at least one dose of study drug
Groups:
- ABBV-444: Participants administered 1-2 drops of ABBV-444 in each eye as needed, but minimally twice a day for 30 days.
Arm/Group | ABBV-444
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.7 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 38
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 38
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Day 30 in Ocular Surface Disease Index (OSDI) Score
Description: The OSDI is a 12-question survey for participants to document their dry eye disease symptoms. The OSDI consists of a 5-point scale ranging from 0 (none of the time) to 4 (all of the time), with higher scores representing greater disability. The scores from the 12 questions are totaled and converted to an overall score ranging from 0 (no disability) to 100 (complete disability). A negative number change from baseline represents an improvement.
Time Frame: Baseline to Day 30
Population: The analysis is based on the full analysis set (FAS), consisting of all participants who were eligible based on the inclusion and exclusion criteria and completed 30 days of treatment for this study.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- ABBV-444: Participants administered 1-2 drops of ABBV-444 in each eye as needed but minimally twice a day for 30 days.
Arm/Group | ABBV-444
Number analyzed (Participants) | 34
score on a scale | -6.8 (15.0)

2. Secondary Outcome: Patient Eye Drop Experience (PEDE) Survey Scores at Day 30 (Visual Analog Scale)
Description: The PEDE Survey is a 13-item questionnaire that evaluates the short- and long-term subjective experience in comfort and vision as well as tolerability, using a scale ranging from 0 (strongly disagree) to 100 (strongly agree). On Day 30, participants were asked to retrospectively recall their experiences after 5 minutes, 30 minutes, 24 hours, and 5 days of when they administered the eye drops
Time Frame: Day 30
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ABBV-444
Number analyzed (Participants) | 34
score on a scale
  The study eye drops do not cause stinging or burning in my eyes (5 minutes) | 76.4 (36.7)
  Study eye drops provided immediate relief of my eye dryness when putting in my eyes (5 minutes) | 77.1 (27.9)
  Study eye drops immediately soothed my eye dryness when putting in my eyes (5 minutes) | 81.3 (25.3)
  Did not experience much blurry/fluctuating vision after putting study eye drops in my eyes (5 mins) | 77.5 (30.4)
  Study eye drops provided immediate comfort to my eye dryness when putting in my eyes (5 minutes) | 84.1 (21.1)
  The study eye drops are very soothing for my eye dryness (30 minutes) | 82.0 (25.6)
  The study eye drops did not feel sticky (30 minutes) | 78.6 (30.8)
  The study eye drops continued to provide relief of my eye discomfort (30 minutes) | 84.6 (20.7)
  The study eye drops continued to provide comfort to my eye dryness (30 minutes) | 85.7 (21.0)
  The study eye drops provided relief of my eye dryness day and night (24 hours) | 84.4 (20.0)
  The study eye drops provided comfort to my eye dryness day and night (24 hours) | 84.5 (21.5)
  The study eye drops provided lasting relief of my eye dryness (5 days) | 83.8 (23.2)
  The study eye drops have provided relief during conditions that lead to eye dryness (5 days) | 82.0 (22.6)

3. Secondary Outcome: Change From Baseline in Symptom Scores (Visual Analog Scale) Within 5 Minutes Post Administration of ABBV-444
Description: The Current Symptom Survey is a 5-item questionnaire where the participants rate their ocular symptoms at the present moment using a scale ranging from 0 (strongly disagree) to 100 (strongly agree). Surveys were completed 5 minutes following the first administration of study eye drops. A negative number change from baseline represents an improvement.
Time Frame: Baseline (T0) to 5 minutes (T5)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ABBV-444
Number analyzed (Participants) | 34
score on a scale | -10.1 (10.6)

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse event tables include events reported from enrollment to end of study. Safety events (per protocol) were collected from enrollment through the 30 day treatment period.
Arm/Group | ABBV-444
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-02): https://cdn.clinicaltrials.gov/large-docs/67/NCT05878067/Prot_SAP_000.pdf